CLINICAL TRIAL: NCT02593838
Title: Diagnostic Value and Practicability of Dynamic CT Stress and Rest Myocardial Perfusion Imaging in Daily Clinical Practice - A Monocentric Prospective Diagnostic Study
Brief Title: Dynamic CT Myocardial Perfusion Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USZ-2015-0393
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTP and SPECT-MPI (Other): Every patient enrolled will undergo CT-MPI and SPECT-MPI. The latter is clinically indicated,.
  Interventions: Other: CT-MPI and SPECT-MPI

INTERVENTIONS:
Other: CT-MPI and SPECT-MPI — All patients undergo CT-MPI plus SPECT-MPI

SUMMARY:
This study aims at evaluating the feasibility of CT myocardial perfusion imaging in daily clinical practice and compare it to SPECT perfusion imaging in order to assess sensitivity and specifity of CT myocardial perfusion imaging compared to SPECT.

DETAILED DESCRIPTION:
If after the clinically indicated CCTA a myocardial perfusion examination is indicated, first a single ultra low dose CT scan will be performed to look for late enhancement of potentially scarred myocardium. Together with the contrast agent co-injection of the clinically indicated tracer 99mTc-Tetrofosmin will be performed for later scintigraphic perfusion evaluation. After stress perfusion imaging CT rest perfusion imaging will be performed in a similar fashion. After acquisition of CT rest perfusion images scintigraphic stress and rest image acquisition will be performed as in daily clinical routine with an additional administration of 99mTc-Tetrofosmin resting dose if necessary.

CT stress and rest perfusion will be compared to the clinically indicated and well established SPECT examination.

ELIGIBILITY:
Inclusion Criteria:

* Referral for cardiac hybrid imaging with CCTA and SPECT
* Male and Female subjects 18 years of age or older,
* Written informed consent by the participant after information about the project

Exclusion Criteria:

* Contraindications for CCTA (including renal failure with a GFR <60ml/min/1.73m2, allergies to ionidated constrast agents)
* Inability to follow the examination procedure due to language barriers, mental disease, dementia etc.
* Pregnancy or breast feeding
* Known allergies to iodinated contrast agent (Visipaque ®), 99mTc-Tetrofosmin (Myoview ®), betablockers (Beloc i.v. ®) or nitrates (Isoket -Spray®)
* Hypersensitivity to adenosine
* Asthma bronchiale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-09; Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Validation of CT-MPI against SPECT-MPI | 2 years
  Sensitivity and specificity of CT-MPI to diagnose obstructive coronary artery disease using SPECTR-MPI as the standard reference

SECONDARY OUTCOMES:
Parameters influencing image quality of CT-MPI - Body physique | 2 years
  Correlation between visually assessed image quality of CT-MPI and patient's body mass index
Parameters influencing image quality of CT-MPI - Heart rate | 2 years
  Correlation between visually assessed image quality of CT-MPI and patient's heart rate during the scan

CONTACTS AND LOCATIONS:
Overall Officials: Ronny R Buechel, MD, Principal Investigator — University Hospital Zurich, Department of Nuclear Medicine
Locations (1):
- Department of Nuclear Medicine, University Hospital Zurich, Zurich, Switzerland